CLINICAL TRIAL: NCT05136677
Title: A Phase II, Randomized, Open-label Trial of Nivolumab in Combination With Ipilimumab Versus Pemetrexed With Cisplatin or Carboplatin as First-line Therapy for Unresectable Pleural Mesothelioma in Chinese Participants
Brief Title: A Study to Evaluate Nivolumab in Combination With Ipilimumab Versus Pemetrexed With Cisplatin or Carboplatin for Unresectable Pleural Mesothelioma in Chinese Participants
Acronym: CheckMate 6DW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-6DW; U1111-1265-3913 (Other: WHO)
Record Dates: First submitted 2021-11-18; First posted 2021-11-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mesothelioma, Malignant
Keywords: Malignant Pleural Mesothelioma (MPM); Nivolumab; Ipilimumab
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Nivolumab; Ipilimumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm B (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Arm A
Biological: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy
  Arms: Arm A
Drug: Pemetrexed — Specified dose on specified days
  Arms: Arm B
Drug: Cisplatin — Specified dose on specified days
  Arms: Arm B
Drug: Carboplatin — Specified dose on specified days
  Arms: Arm B

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the combination of nivolumab and ipilimumab in Chinese participants with malignant pleural mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of Malignant Pleural Mesothelioma (MPM) with determination of epithelioid vs non-epithelioid histology
* Must have advanced unresectable disease that is not amenable to therapy with curative intent (surgery with or without chemotherapy)
* Available tumor samples for centralized testing
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Measurable disease

Exclusion Criteria:

* Primitive peritoneal, pericardial, testis or tunica vaginalis mesothelioma
* Brain metastasis, except if surgically resected or treated with stereotaxic radiotherapy
* Prior therapy for MPM (including chemotherapy, radical pleuropneumonectomy and non-palliative radiotherapy)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 58 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by modified Response Evaluation Criteria in Solid Tumors (m-RECIST) by Investigator | Up to 58 months
Progression Free Survival (PFS) by m-RECIST by Investigator | Up to 58 months
Incidence of Adverse Events (AEs) | Up to 58 months
Incidence of Serious Adverse Events (SAEs) | Up to 58 months
Incidence of immune-related AEs | Up to 58 months
Incidence of deaths | Up to 58 months
Incidence of participants with laboratory abnormalities | Up to 58 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- China (21):
  - Local Institution - 0009, Beijing, Beijing Municipality
  - Local Institution - 0013, Harbin, Heilongjiang
  - Local Institution - 0006, Zhengzhou, Henan
  - Local Institution - 0005, Changsha, Hunan
  - Local Institution - 0023, Wuhan, Hunan
  - Local Institution - 0015, Yangzhou, Jiangsu
  - Local Institution - 0003, Changchun, Jilin
  - Local Institution - 0004, Shenyang, Liaoning
  - Local Institution - 0021, Shenyang, Liaoning
  - Local Institution - 0037, Jinan, Shandong
  - Local Institution - 0030, Qingdao, Shandong
  - Local Institution - 0001, Shanghai, Shanghai Municipality
  - Local Institution - 0033, Taiyuan, Shanxi
  - Local Institution - 0029, Chengdu, Sichuan
  - Local Institution - 0007, Tianjin, Tianjin Municipality
  - Local Institution - 0018, Tianjin, Tianjin Municipality
  - Local Institution - 0010, Kunming, Yunnan
  - Local Institution - 0014, Hangzhou, Zhejiang
  - Local Institution - 0020, Hangzhou, Zhejiang
  - Local Institution - 0012, Ningbo, Zhejiang
  - Local Institution - 0016, Ningbo, Zhejiang

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com